CLINICAL TRIAL: NCT07313969
Title: The Impact of Ultra-Low-Flow Sevoflurane Anesthesia on Carbon Footprint and Cost: A Randomized Controlled Study in Cardiac Surgery Patients
Brief Title: Ultra-Low-Flow Anesthesia and Carbon Footprint
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Collaborators: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Ekin Guran, MD, consultant anesthesiologist, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ultra_low_flow
Record Dates: First submitted 2025-12-10; First posted 2026-01-02 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-12

CONDITIONS: Low Flow Anesthesia; Sevoflurane Anesthesia; Cardiac Surgery
Keywords: low flow anesthesia; ultra low flow anesthesia; carbon footprint

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and postoperative outcome assessors will be blinded to group allocation. The anesthesia provider cannot be blinded due to visible gas flow settings; however, they will not be involved in postoperative data collection or analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultra-Low-Flow Group (0.5 L/min) (Active Comparator): Sevoflurane anesthesia with fresh gas flow maintained at 0.5 L/min throughout the maintenance period. A 2 lt/min fresh gas flow will be used in the preoxygenation and intubation phase.
  General anesthesia will be maintained with sevoflurane at a fresh gas flow rate of 0.5 L/min using an oxygen and air mixture. The flow rate will be kept constant from post-induction stabilization until the end of the surgery. Ventilation will be paused during cardiopulmonary bypass.
  Interventions: Drug: ultra low flow anesthesia
- Normal-Flow Group (2.0 L/min) (Active Comparator): Sevoflurane anesthesia with fresh gas flow maintained at 2.0 L/min throughout maintenance period. The flow rate will be kept constant from post-induction stabilization until the end of surgery. Ventilation will be paused during cardiopulmonary bypass
  Interventions: Drug: normal flow anesthesia

INTERVENTIONS:
Drug: ultra low flow anesthesia — General anesthesia will be maintained with sevoflurane at a fresh gas flow rate of 0.5 L/min using oxygen and air mixture. The flow rate will be kept constant from post-induction stabilization until the end of cardiopulmonary bypass.
  Arms: Ultra-Low-Flow Group (0.5 L/min)
Drug: normal flow anesthesia — General anesthesia will be maintained with sevoflurane at a fresh gas flow rate of 2.0 L/min using oxygen and air mixture. The flow rate will be kept constant from post-induction stabilization until the end of cardiopulmonary bypass.
  Arms: Normal-Flow Group (2.0 L/min)

SUMMARY:
This is a prospective, randomized controlled clinical trial evaluating the effects of ultra-low fresh gas flow (0.5 L/min) versus normal fresh gas flow (2.0 L/min) sevoflurane anesthesia in adult patients undergoing on-pump cardiac surgery. The study aims to determine whether ultra-low-flow anesthesia can be used safely to reduce volatile anesthetic consumption and environmental emissions without compromising hemodynamic stability or anesthetic depth.

Eligible adult patients scheduled for elective coronary artery bypass grafting (CABG) or valve surgery under general anesthesia will be randomized in a 1:1 ratio to one of two groups: ultra-low-flow (0.5 L/min) or normal-flow (2.0 L/min). All other anesthetic techniques, including induction drugs, ventilation parameters, temperature management, and perfusion strategies, will be standardized.

The primary outcome is the total amount of sevoflurane consumed per case. Secondary outcomes include intraoperative hemodynamic parameters (heart rate, mean arterial pressure), depth of anesthesia (BIS/MAC values), postoperative recovery times, and estimated carbon dioxide equivalent (CO₂e) emissions.

Outcome assessors and data analysts will remain blinded to group allocation. The findings of this study are expected to provide new evidence regarding the safety, efficiency, and environmental benefits of ultra-low-flow anesthesia techniques in cardiac surgery.

DETAILED DESCRIPTION:
This randomized controlled trial investigates the impact of ultra-low-flow (0.5 L/min) versus normal-flow (2.0 L/min) sevoflurane anesthesia on anesthetic consumption, intraoperative hemodynamics, and environmental footprint during on-pump cardiac surgery. Although low-flow anesthesia is known to reduce anesthetic agent use and greenhouse gas emissions, evidence regarding its safety and efficiency during cardiopulmonary bypass procedures remains limited.

Adult patients scheduled for elective CABG or valve surgery will be randomly assigned to either an ultra-low-flow or normal-flow group. Randomization will be performed using a computer-generated sequence with variable block sizes and allocation concealment via sequentially numbered, opaque, sealed envelopes. All participants will receive standardized induction, perfusion, and maintenance techniques according to institutional cardiac anesthesia protocols.

The primary outcome measure is total sevoflurane consumption per patient, assessed through vaporizer readings and anesthetic gas analyzer data. Secondary outcomes include intraoperative mean arterial pressure, heart rate, BIS/MAC values, body temperature, recovery characteristics, and calculated CO₂ equivalent emissions. Outcome assessors and data analysts will remain blinded to group allocation.

This study is designed to evaluate both clinical and ecological aspects of anesthetic practice. It aims to determine whether ultra-low-flow anesthesia can provide equivalent anesthetic quality while offering substantial reductions in agent consumption and environmental impact. The findings may contribute to establishing safer and more sustainable anesthesia standards for cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18-80 years
* Scheduled for elective on-pump CABG or valve surgery
* ASA physical status II-III
* Written informed consent obtained

Exclusion Criteria:

* Emergency surgery
* Severe hepatic or renal dysfunction
* Known allergy to volatile anesthetics
* Significant pulmonary disease (e.g., COPD with GOLD III-IV)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2025-07-30 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2026-01-15 (Actual)

PRIMARY OUTCOMES:
Total sevoflurane consumption (mL per case), measured at the end of surgery. | throughout the surgery

SECONDARY OUTCOMES:
carbon footprint | throughout the surgery
  Estimated CO₂e emissions (calculated from anesthetic use)

CONTACTS AND LOCATIONS:
Locations (1):
- Etlik City Hospital, Ankara, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] McGain F, Sheridan N, Wickramarachchi K, Yates S, Chan B, McAlister S. Carbon Footprint of General, Regional, and Combined Anesthesia for Total Knee Replacements. Anesthesiology. 2021 Dec 1;135(6):976-991. doi: 10.1097/ALN.0000000000003967. PMID 34529033